CLINICAL TRIAL: NCT04495140
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD STUDY IN HEALTHY ADULT MALE PARTICIPANTS TO ASSESS THE MASS BALANCE, ABSOLUTE BIOAVAILABILITY, FRACTION ABSORBED, AND PHARMACOKINETICS OF [14C]PF-06882961
Brief Title: Study To Characterize Mass Balance, Absolute Bioavailability, Fraction Absorbed And Pharmacokinetics Of 14C PF-06882961
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C3421009; 2019-002584-10 (EudraCT Number)
Record Dates: First submitted 2020-07-16; First posted 2020-07-31 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteer
Keywords: bioavailability; excretion; metabolism; absorption
MeSH Terms: interventions — danuglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral [14C]PF-06882961, 50 mg (Experimental): In this arm, a single oral dose of [14C]PF-06882961, 50 mg will be administered as a liquid formulation.
  Interventions: Drug: [14C]PF-06882961, 50 mg
- Oral PF-06882961 50 mg and intravenous [14C]PF-06882961 100 ug (Experimental): In this arm, single oral dose of unlabeled PF-06882961, 50 mg will be administered as a liquid formulation. Approximately 3 hours after the administration of the unlabeled oral dose, a single dose of [14C]PF-06882961, 100 ug, will be administered via intravenous infusion.
  Interventions: Drug: PF-06882961, 50 mg and [14C]PF-06882961, 100 ug

INTERVENTIONS:
Drug: [14C]PF-06882961, 50 mg — A single oral dose of [14C]PF-06882961, will be administered as a liquid formulation.
  Arms: Oral [14C]PF-06882961, 50 mg
Drug: PF-06882961, 50 mg and [14C]PF-06882961, 100 ug — A single, oral, unlabeled dose of PF-06882961, 50 mg will be administered as a liquid formulation. Approximately 3 hours after the administration of the unlabeled oral dose, a single dose of [14C]PF-06882961 will be administered via intravenous infusion.
  Arms: Oral PF-06882961 50 mg and intravenous [14C]PF-06882961 100 ug

SUMMARY:
This study is a Phase 1, open-label, non-randomized, 2-period, fixed sequence study to characterize the metabolic profile and routes of excretion of oral [14C]PF-06882961 and to evaluate the absolute oral bioavailability of PF-06882961 and fraction absorbed of [14C]PF-06882961 in reference to intravenous [14C]PF-06882961 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Male participants between 18 to 54 years of age
* Healthy and capable of signing informed consent document
* Willing to comply to all scheduled visits, lab tests, lifestyle considerations and study procedures
* Body mass index (BMI) of 17.5 to 30 kg/m2; and a total body weight ≥50 kg (110 lb).

Exclusion Criteria:

* acute or chronic medical or psychiatric condition including recent (within the past year)
* Surgical procedures like gastrectomy, cholecystectomy, Irregularity in bowel movements
* Use of prescription or non-prescription drugs and dietary and herbal supplements within 14 days prior to the first dose of investigational product.
* Previous administration with an investigational drug within 60 days (or as determined by the local requirement) preceding the first dose of investigational product used in this study.
* Known prior participation in a trial involving PF-06882961 or known intolerance to a GLP-1R agonist.
* A positive urine drug test on screening or Day -1.
* Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* Participants with abnormalities in clinical laboratory tests including ECGs, vital signs, liver function tests, myocardial infarction
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb). Hepatitis B vaccination is allowed.
* History of alcohol or tobacco abuse or binge drinking and/or any other illicit drug use or dependence within past 6 months.
* Subjects whose occupation requires exposure to radiation or monitoring of radiation exposure.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia only if heparin is planned to flush intravenous catheters.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Total recovery of radioactivity in urine and feces, following oral administration of [14C] PF-06882961 in period 1 | Baseline through approximately hour 312 (day 14). Period 1 is 14 days
  Total recovery of radioactivity in urine and feces, and both routes combined, expressed as a percent of total oral radioactive dose administered.

SECONDARY OUTCOMES:
Metabolite profiling/identification in plasma, urine, and feces | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96-312 hour (hr)
  Metabolic profiling/identification and determination of relative abundance of [14C]PF-06882961 and the metabolites of [14C]PF-06882961 in plasma, urine, and feces.
Plasma Cmax to describe plasma PK of total radioactivity following administration of single, oral dose of [14C] PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Maximum Observed Plasma Radioactivity
Plasma Tmax to describe the PK of total radioactivity following administration of single, oral dose of [14C]PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Time to Reach Maximum Observed Plasma Radioactivity
Plasma AUClast to describe PK of total radioactivity following administration of single, oral dose of [14C] PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Area under the plasma radioactivity-time profile from time 0 to time of the last quantifiable concentration (Clast)
Plasma AUCinf to describe plasma PK of total radioactivity following administration of single, oral dose of [14C] PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  AUCinf is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Plasma elimination t½ to describe plasma PK of total radioactivity following administration of single, oral dose of [14C] PF-06882961 | 00, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Plasma elimination half-life is the time measured for the plasma radioactivity to decrease by one half.
Plasma Cmax to describe the plasma PK of PF-06882961 following administration of single, oral dose of [14C] PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Maximum Observed Plasma Concentration
Plasma Tmax to describe the plasma PK of PF-06882961 following administration of single, oral dose of [14C]PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Time to Reach Maximum Observed Plasma Concentration
Plasma AUClast to describe PK of PF-06882961 following administration of single, oral dose of [14C] PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Area under the plasma concentration-time profile from time 0 to time of the last quantifiable concentration (Clast)
Plasma AUCinf to describe plasma PK of PF-06882961 following administration of single, oral dose of [14C] PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  AUCinf is Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Mean residence Time (MRT )following administration of a single, intravenous dose of [14C]PF 06882961 | 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72 hr
  where MRT is the Mean Residence Time
Systemic Clearance (CL) following administration of a single, intravenous dose of [14C]PF 06882961 | 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72 hr
  Systemic clearance, CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Volume of distribution at steady state (Vss) following administration of a single, intravenous dose of [14C]PF 06882961 | 0, 1, 2, 4, 5, 6, 8, 10, 12, 24, 36, 48, 72 hr
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state.
Absolute oral bioavailability (F) | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Absolute oral bioavailability following administration of a single oral dose of PF-06882961 in reference to a single intravenous dose of [14C]PF-06882961
Fraction of dose absorbed following single oral administration of [14C]PF-06882961 | 0, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96-312hr
  Fraction absorbed calculated from ratio of total urinary radioactivity following oral administration in reference to intravenous administration
Number of participants with adverse events | Baseline in Period 1 up to 32 days after the period 2 doses, for a total of approximately 46 days
  adverse events
Plasma elimination t½ to describe plasma PK of PF-06882961 following administration of single, oral dose of [14C] PF-06882961 | 00, 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hr
  Plasma elimination half-life is the time measured for the plasma radioactivity to decrease by one half.
Number of participants with safety laboratory test results above/below certain threshold | baseline, day 5-14 of period 1 (period 1 is 14 days), day 3-8 of period 2 (period 2 is 8 days)
  lab tests
Number of participants with ECG measurements above/below certain threshold | baseline, day 5-14 of period 1 (period 1 is 14 days), day 3-8 of period 2 (period 2 is 8 days)
  ECGs
Number of participants with vital measurements above/below certain threshold | baseline, day 5-14 of period 1 (period 1 is 14 days), day 3-8 of period 2 (period 2 is 8 days)
  vitals

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Netherlands (2):
  - PRA Health Sciences, Groningen
  - PRA Health Sciences Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3421009